CLINICAL TRIAL: NCT02193334
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of Intrathecal Injection of KP-100IT in Subjects With Acute Spinal Cord Injury
Brief Title: Phase I/II Study of KP-100IT in Acute Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kringle Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KP-100-ND002
Record Dates: First submitted 2014-06-27; First posted 2014-07-17 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Spinal Cord Injuries
Keywords: Hepatocyte Growth Factor; HGF; KP-100IT; Intrathecal injection
MeSH Terms: conditions — Spinal Cord Injuries; Deafness, Autosomal Recessive 39 | interventions — Hepatocyte Growth Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KP-100IT (Active Comparator): Intrathecal injection of 0.6 mg HGF starting at 72 hours since the injury and repeating weekly 5 times
  Interventions: Drug: KP-100IT
- Placebo (Placebo Comparator): Intrathecal injection of placebo starting at 72 hours since the injury and repeating weekly 5 times
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KP-100IT
  Other Names: Hepatocyte Growth Factor; HGF
  Arms: KP-100IT
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is randomized, double-blind, placebo-controlled Phase I/II study designed to evaluate safety and efficacy of KP-100IT, code of Hepatocyte Growth Factor (HGF) formulation for intrathecal injection, as a treatment for acute spinal cord injury. The study is conducted at two clinical sites in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years and equal to or less than 75 years
* Cervical spinal cord injury, and Grade A, B1 or B2 in the modified Frankel Scale at 72 hours since the injury
* Subjects able to provide written informed concent, which may require a relative to sign if arm/hand function of the subject is compromised

Exclusion Criteria:

* Spinal cord injury at C1-C2 0r C2-C3 level
* Patients not to able to start rehabilitation within a week by setup of respirator or other reason
* First dose of the study drug will not be given within 78 hours since the injury
* History of spinal cord injury or abnormality in spinal cavity. Or current considerable meningeal damage
* Outcome assessment will not be conducted adequately through damage on injuries other than the injury
* High-dose steroid therapy within 30 days before the entry
* Patients who have diseases such as serious liver disorder, renal disorder, hear disease, blood dyscrasia, metabolism disorder and infections
* History of malignant tumor
* Patients who participated in other clinical study within 30 days before the entry
* Patients who have allergies to drug scheduled to be used in the study
* Administration of the study drug to the area of spinal cord injury is not appropriate for example by intrathecal infections or intrathecal tumor
* Patients not able to understand "informed consent" properly
* Patients who are nursing or may be pregnant
* Investigator considers that the patient is not appropriate for participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Number and degree of adverse events | 24 weeks
  Adverse events will be judged by general condition, vital sign, electrocardiogram, MRI, blood chemistry, hematology, urinalysis, cerebrospinal fluid examination, and antibody formation
Change of ASIA (American Spinal Injury Association) motor score from baseline at 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Change of ASIA motor score from baseline at 12 weeks | 12 weeks
Time-dependent change of ASIA motor score from baseline | 24 weeks
Time-dependent change of ASIA sensory score from baseline | 24 weeks
Time-dependent grade change of modified Frankel scale from baseline | 24 weeks
Time-dependent change of P-100 concentration in plasma and cerebrospinal fluid | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Etsuro HASHIMURA, Study Director — Kringle Pharma, Inc.
Locations (2):
- Japan (2):
  - Spinal Injuries Center, Iizuka, Fukuoka
  - Hokkaido Chuo Rosai Hospital Sekison Center, Bibai, Hokkaido